CLINICAL TRIAL: NCT03034590
Title: How to Identify Fatigue in Stroke Patients: Validity of the Post-stroke Fatigue Case Definition
Brief Title: How to Identify Fatigue in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Karsten Overgaard, MD, Herlev Hospital
Other Study IDs: ID 3-3013-583/1/
Record Dates: First submitted 2016-10-12; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Post Stroke Fatigue; Stroke
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire

SUMMARY:
This study will translate an English case definition of poststroke fatigue and validate it against the Multidimensional Fatigue Questionnaire-20 and the Fatigue Severity Scale

ELIGIBILITY:
Inclusion Criteria:

Patients with a clinical stroke within the last 6 months as judged by a senior doctor or by the research assistant.

Patients that have given written informed consent

-

Exclusion Criteria:

Patients with aphasia, dementia or cognitive deficits so severe that they are unable to understand the purpose of the interview and the questionnaire. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients with a new stroke within 120 days
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean MFI-20 score for case positive patients | at inclusion in the trial
  Describes validity of the case definition with regards to the MFI-20 questionnaire
Mean FSS-7 score for case positive patients | At inclusion in the trial
  Describes validity of the case definition with regards to the FSS-7 questionnaire

SECONDARY OUTCOMES:
inter rater variability of the case definition | within a week
  Reinterview by a second interviewer
Optimal cut off score for case positiveness on MFI-20 and FSS | at inclusion in the trial (which is the time the values used are measured)
  decide the optimal cut-off score on the two questionnaires to define case positiveness

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Overgaard, MD, Principal Investigator — Department of Neurology, Herlev Hospital
Locations (1):
- Department of Neurology, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No